CLINICAL TRIAL: NCT03472768
Title: The Impact of Age-dependent Haptoglobin Deficiency on Plasma Free Hemoglobin Levels During Extracorporeal Membrane Oxygenation Support
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-2058
Record Dates: First submitted 2018-02-02; First posted 2018-03-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Failure
Keywords: ECMO
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECMO-supported group: Thirty critically-ill children (age newborn to 18 years) who are intubated and supported by ECMO. Normal adult-level haptoglobin concentrations are achieved by 6-12 months of age. We will target enrollment of 15 subjects less than 12 months of age and 15 subjects over 12 months of age
  Interventions: Diagnostic Test: Plasma Haptoglobin Concentration
- Age-matched group with respiratory failure: Sixty critically-ill children (age newborn to 18 years) who are intubated with acute respiratory failure due to any cause and not supported by ECMO. Two control subjects will be enrolled for every 1 experimental ECMO subject.
  Interventions: Diagnostic Test: Plasma Haptoglobin Concentration

INTERVENTIONS:
Diagnostic Test: Plasma Haptoglobin Concentration — N/A, comparison of haptoglobin concentration between groups

SUMMARY:
Newborns and children with life-threatening heart and lung failure may require support with ECMO (extracorporeal membrane oxygenation). With ECMO, oxygen and carbon dioxide are exchanged and circulated throughout the body even if the heart is unable to do so. Unfortunately, ECMO can cause breakdown of the red blood cells (known as hemolysis). For unclear reasons, newborns are at particularly high risk of hemolysis while being supported by ECMO. The amount of hemolysis is measured with concentrations of a breakdown product from red blood cells known as free hemoglobin. One possible reason for high free hemoglobin levels in newborns on ECMO could be related to another blood protein called haptoglobin. Haptoglobin is known to help in clearing free hemoglobin through the kidneys into the urine. However, haptoglobin levels in newborns can be very low and increases slowly during the first few months of life. Free hemoglobin may be inappropriately high in newborns supported by ECMO because of low levels of haptoglobin. The purpose of this study is to characterize haptoglobin, free hemoglobin, and hemolysis in newborns and children supported by ECMO and compare those values to age-matched newborns and children not on ECMO.

ELIGIBILITY:
Inclusion Criteria:

* ECMO group - Thirty critically-ill children (age newborn to 18 years) who are intubated and supported by ECMO. We will target enrollment of 15 subjects less than 12 months of age (with at least 10 subjects enrolled less than 6 months of age) and 15 subjects over 12 months of age. These targets are set to address the secondary aim in the context of normal adult-level haptoglobin concentrations reportedly achieved by 6-12 months of age.
* Age-matched control group - Sixty critically-ill children (age newborn to 18 years) who are intubated with acute respiratory failure due to any cause and not supported by ECMO. Two control subjects will be enrolled for every 1 experimental ECMO subject. Age-matching will be performed by the following age groups:

  * Neonates 37-40 weeks gestation
  * Neonates 40-42 weeks gestation
  * Neonates 42-44 weeks gestation
  * Neonates 44-46 weeks gestation
  * Neonates 46-48 weeks gestation
  * Infants 2-4 months of age
  * Infants 4-6 months of age
  * Infants 6-12 months of age
  * Children 1-4 years of age
  * Children 4-8 years of age
  * Children 8-12 years of age
  * Children 12-18 years of age

Age-matched control subjects will proceed through the 3 total blood sample collections even if endotracheal extubation occurs within the 3 days of study participation. Age-matching is intended to collect a sample population comparable to the ECMO subject population. We will not match to gender.

Exclusion Criteria (both groups, ECMO and age-matched controls):

* Personal or family history of thrombotic, hemorrhagic, or hemolytic disease.
* Personal history of hematologic malignancy.
* Premature neonates less than 37-weeks gestation and/or less than 2 kg in weight.
* Infection will not be an excluding factor for either subject group.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically-ill children with respiratory failure requiring mechanical circulatory and/or respiratory support.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Characterize the relationship between plasma haptoglobin and free hemoglobin levels in children supported by ECMO. | Daily for 7 days
  Serum Haptoglobin (Hp) will be measured daily for 7 days in subjects supported by Extracorporeal Membrane Oxygenation (ECMO). In particular, the relative deficiency of Hp production in neonates will be associated with higher Hp levels. In older children with normal and adequate Hp production, there will be consistently low fHgb concentrations regardless of the other risk factors for hemolysis during ECMO support.
Characterize the relationship between plasma haptoglobin and free hemoglobin levels in children supported by ECMO. | 7 days
  Plasma free hemoglobin (fHgb) concentrations will be extracted from the medical record. Periods of high fHgb associated with hemolysis during ECMO support will be associated with deficiency of Hp at that time.

SECONDARY OUTCOMES:
Characterize the deficiency of plasma haptoglobin at birth. | Daily for 3 days
  Serum Hp and fHgb will be measured daily for 3 days in age-matched control subjects to characterize levels in a cohort of critically-ill children comparable to the ECMO cohort. Neonates and children with non-ECMO supported critical illness will have negligible risk for hemolysis and, thus, low plasma fHgb. Serum Hp concentrations will be similar to the previously-characterized norms in healthy subjects (eg. deficient at birth until 6-12 months of age).

CONTACTS AND LOCATIONS:
Overall Officials: John Kim, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado and the University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided